CLINICAL TRIAL: NCT04118153
Title: Early Markers of Disease and Response to Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sandra Lord, MD (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Medical College of Wisconsin (Other)
Responsible Party: Sponsor-Investigator, Sandra Lord, MD, Clinical Director, Center for Interventional Immunology, Benaroya Research Institute
Organization: Benaroya Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DREAMT V1.0
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Abatacept

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abatacept (Experimental): Abatacept will be given by a subcutaneous (SC) formulation weekly for three months.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Abatacept will be administered by subcutaneous injections weekly for 3 months. Dosing is according to body weight at screening visit and will be administered as follows: up to 25 kg receive 50 mg (0.4 mL); 25 to <50 kg receive 87.5 mg (0.7 mL), and > 50 kg receive 125 mg (1.0 mL) per dose.
  Other Names: ORENCIA

SUMMARY:
The purpose of this study is to identify early immune markers associated with response to treatment with abatacept in individuals with Type 1 diabetes (T1D). In this open label mechanistic study, participants who were recently diagnosed with T1D (males or females, ages 6-45 and <7months from T1D diagnosis) will be treated with a short-course of abatacept (weekly subcutaneous injections for 3 months). Participants will undergo baseline and repeated mixed meal tolerance testing (MMTT) to assess disease progression and blood samples will be obtained at frequent intervals to measure changes in immune markers.

ELIGIBILITY:
Inclusion Criteria:

1. ≤ 7 months from type 1 diabetes diagnosis based on ADA criteria
2. > 21 days from type 1 diabetes diagnosis or metabolically stable per study physician assessment
3. Males and females 6-55 years of age, inclusive, at time of screening visit
4. Peak MMTT stimulated C-peptide ≥ 0.2 pmol/ml
5. Females of child-bearing age must be willing to use effective birth control for 1 year (which may include abstinence) from screening visit and undergo regular pregnancy testing
6. Up to date for clinically recommended immunizations prior to screening
7. Willing to forgo live vaccines 3 months prior to the screening visit until three months following last study drug administration
8. Willing and able to give informed consent or have parent or legal guardian provide informed consent if the subject is < 18 years of age
9. Weight ≥ 20 kg at baseline visit
10. HbA1c ≤ 8.5% at baseline visit
11. Positive for at least 1 diabetes autoantibody (excluding mIAA in those who have received ≥ 2 weeks of exogenous insulin therapy)

Exclusion Criteria:

1. Concurrent or recent (within the past 30 days of screening MMTT (visit -1)) use of non-insulin therapies aimed to control hyperglycemia
2. Females who are pregnant or lactating
3. Immunodeficiency or clinically significant chronic lymphopenia
4. Have an active infection at time of screening or baseline visit
5. Recent exposure, or possible or known active SARS-CoV-2 infection as defined by public health guidelines
6. Positive QuantiFERON or PPD TB test, history of tuberculosis, or active TB infection
7. Active infection with EBV or CMV, defined by real-time PCR
8. History of other clinically significant autoimmune disease needing chronic therapy with biologics or steroids with the exception of celiac disease and stable thyroid disease
9. Require use of other immunosuppressive agents for any other condition
10. Use of medications known to influence glucose tolerance
11. Have any complicating medical or psychological issues or abnormal clinical laboratory results that interfere with study conduct or cause increased risk. These include pre-existing cardiac disease, COPD, neurological, or clinically significant blood count abnormalities (such as lymphopenia, leukopenia, or thrombocytopenia).
12. Have serologic evidence of current or past HIV, Hepatitis B (positive for Hepatitis B core antibody or surface antigen), or Hepatitis C infection.
13. Have a history of malignancies
14. Receipt of live vaccine (MMR, intranasal influenza, varicella, rotatvirus) in 3 months before treatment

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Change in insulin antibody titers (NIDDK units/mL) | 0 to 2 weeks
  Insulin antibody titers
Change in frequency of B cells within total PBMC (%) | 0 to 2 weeks
  % of B cells
Change in inflammatory Index by serum transcriptional exposure assay (composite score) | 0 to 2 weeks
  Inflammatory Index (359). This is an inflammatory index based on transcription of 359 probe sets (I.I.359) calculated by dividing the average signal intensity of the 103 probe sets generally annotated as 'inflammatory' by the average signal intensity of the 256 probe sets generally annotated as 'regulatory'
Change in B-cell transcriptional module (CD19.mod) (composite score) | 0 to 2 weeks
  CD19 mod is composite score of B cell transcripts.
Change in islet-specific exhausted CD8 T cells (%) | 0 to 2 weeks
  % of CD8+ T cells (CD8+PD-1+KLRG1+CD57-)
Change in EOMES CD8 whole blood gene expression signature (composite score) | 0 to 2 weeks
  Gene transcript score for EOMES module
Change in frequency of TfH within total CD4 T cells (%) | 0 to 2 weeks
  % of TfH cells within CD4+ T cells

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Principal Investigator — Benaroya Research Institute at Virginia Mason
Locations (2):
- United States (2):
  - Benaroya Research Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No